CLINICAL TRIAL: NCT03952689
Title: Automatic Urine Output Measuring Device Performance Validation and Efficacy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-19-5839-ER-CTIL
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Urine Output Decreased
MeSH Terms: conditions — Oliguria

STUDY DESIGN:
Intervention Model Description: Prospective Observational, single arm test, self-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post cardiac surgery patients (Experimental): For all patients, readings of the urine output from both the Serenno system and the collection bag (urinometer) (by camera) will be recorder every 10 minutes, for the duration of 24 hours.
  Interventions: Device: Serenno Medical Automatic Urine Output measuring device

INTERVENTIONS:
Device: Serenno Medical Automatic Urine Output measuring device — Device that measures ongoing urine output will be connecter to the patients catheter. The urine count of the device will be compared to the "gold standard" measurement technique (nurse count).

SUMMARY:
To evaluate the efficacy of Serenno Medical Automatic Urine Output measuring device in patients with indwelling urinary catheter hospitalized in the cardiac surgery intensive care unit.

DETAILED DESCRIPTION:
In order to evaluate the efficacy of Serenno Medical Automatic Urine Output measuring device we will perform a non inferiority of study device in compare with Urinometer (with acceptance of 3% standard deviation), in patients hospitalized in the intensive care unit after cardiac surgery.

Secondary endpoints are to attribute and Identify urine output changes prior to early stage acute renal failure, and identifying urine output changes prior to fluid overload or dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, aged >18 years
* Patients hospitalized in the intensive care unit requiring an indwelling urinary catheter for urine output monitoring for at least 24 hours.

Exclusion Criteria:

* Known urological pathology including but not limited to nephrolithiasis, polycystic kidney disease, congenital abnormalities of the kidneys and or urinary tract, history of obstructive uropathy, advanced chronic kidney disease (stage 4) of any cause.
* Known pregnancy or lactating women.
* Cognitive and/or psychiatric impairment which may not allow cognitive signing on the informed consent unless patient has a legal representative that was appointed prior to patient enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-10-14 (Estimated); Study Completion 2021-10-14 (Estimated)

PRIMARY OUTCOMES:
Urine volume measurement. | 24 hours
  Automatic device urine output measurement in compare with Urinometer

SECONDARY OUTCOMES:
Acute renal failure detection by urine output measurement and creatinine level in the blood. | 24 hours
  To identify urine output changes prior to early stage acute renal failure. Reduction in urine output in hemodynamic stable patients will be followed by creatinine measurement in the blood in order to verify laboratory signs of acute renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Ram, Dr, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No